CLINICAL TRIAL: NCT01422369
Title: Drug-Drug Interaction Study to Assess the Effects of Steady-State Darunavir/Ritonavir on Steady-State Pitavastatin in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction of Darunavir/Ritonavir on Pitavastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NK-104-4.06US
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — pitavastatin; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Subjects (Experimental): pitavastatin 4 mg
  Interventions: Drug: Pitavastatin (NK-104); Drug: Darunavir/Ritonavir (Prezista)

INTERVENTIONS:
Drug: Pitavastatin (NK-104) — Pitavastatin (NK-104) 4mg once daily (QD)
Drug: Darunavir/Ritonavir (Prezista) — Darunavir/Ritonavir (Prezista) 800 mg/100 mg

SUMMARY:
This is a Phase 4, single center, open label, fixed-sequence, multiple dose, 2-way drug-drug interaction study.

DETAILED DESCRIPTION:
This is a Phase 4, single center, open label, fixed-sequence, 2-way drug-drug interaction study.

Each subject will qualify for entry into the study not more than 30 days before admission into the clinical unit. Subjects will check into the clinical unit on Day -1 for baseline assessments. There will be 1 treatment period, with each subject receiving a once daily dose of pitavastatin 4 mg on Days 1 through 5 and Days 12 through 16 and a once daily dose of darunavir/ritonavir 800 mg/100 mg on Days 6 through 16. On Days 1 through 4, 6 through 10, and 12 through 15, study drug will be administered 30 minutes before a standard breakfast. On Days 5, 11, and 16, subjects will fast at least 8 hours before receiving study drug and remain fasted for 4 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteer aged 18 to 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive.
* Subject has normal hematology, serum chemistry, and urinalysis test results
* Subject is able and willing to abstain from alcohol, grapefruit, caffeine or caffeine containing products, St John's wort, and herbal supplements for 4 days before Day 1 and until completion of the study
* Subject is a nonsmoker or has quit smoking at least 6 months before the first dose of study drug and until study completion.

Exclusion Criteria:

* Subject has had any surgery of the gastrointestinal tract likely to affect drug absorption, distribution, metabolism, or excretion.
* Subject has had a previous allergy or intolerance to treatment with pitavastatin, darunavir, ritonavir, sulfonamides, or any drugs in these classes.
* Subject has a history of drug or alcohol abuse.
* Subject has had a clinically significant illness within 4 weeks before the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Morgan, MD, FACS, Study Director — Kowa Research Institute, Inc.
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Yu CY, Campbell SE, Sponseller CA, Small DS, Medlock MM, Morgan RE. Steady-state pharmacokinetics of darunavir/ritonavir and pitavastatin when co-administered to healthy adult volunteers. Clin Drug Investig. 2014 Jul;34(7):475-82. doi: 10.1007/s40261-014-0198-x. PMID 24825411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1st Subject Enrolled 20 April 2011 Last Subject Completed 10 June 2011
Groups:
- All Subjects: All randomized subjects
Period: NK-104 4mg QD
Arm/Group | All Subjects
Started | 28
Completed | 28
Not Completed | 0
Period: Prezista 800mg/100mg QD
Arm/Group | All Subjects
Started | 28
Completed | 28
Not Completed | 0
Period: NK-104 4mg QD & Prezista 800mg/100mg QD
Arm/Group | All Subjects
Started | 28
Completed | 27
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: NK-104 AUC
Time Frame: 16 Days
Population: All subjects with measurable pharmacokinetic (PK) values.
Measure: Mean (Standard Deviation); unit: ng * h/mL
Groups:
- NK-104: NK-104 4mg once daily (QD)
Arm/Group | NK-104
Number analyzed (Participants) | 27
ng * h/mL | 192.00 (80.8)

2. Secondary Outcome: Number of Participants With at Least One Adverse Event.
Time Frame: 16 Days
Population: All subjects who took at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 28
Participants | 2

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 13/28
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=28)
Diarrhea (Gastrointestinal disorders) | 1
Paresthesia (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 2
Feeling cold (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
May not publish.